CLINICAL TRIAL: NCT05869955
Title: A Phase 1, Multicenter, Open-Label Study Of CC-97540 (BMS-986353), CD19-Targeted Nex-T Chimeric Antigen Receptor (CAR) T Cells, in Participants With Severe, Refractory Autoimmune Diseases: Systemic Lupus Erythematosus, Idiopathic Inflammatory Myopathy, Systemic Sclerosis, or Rheumatoid Arthritis (Breakfree-1)
Brief Title: A Study of CC-97540, CD-19-Targeted Nex-T CAR T Cells, in Participants With Severe, Refractory Autoimmune Diseases (Breakfree-1)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Collaborators: Bristol-Myers Squibb Services Unlimited Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA061-1001; 2023-503823-24 (EudraCT Number)
Record Dates: First submitted 2023-05-11; First posted 2023-05-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; Idiopathic Inflammatory Myopathy; Systemic Sclerosis; Rheumatoid Arthritis
Keywords: CC-97540; BMS-986353
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Arthritis, Rheumatoid | interventions — fludarabine; Cyclophosphamide; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-97540 (Experimental)
  Interventions: Drug: CC-97540; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tocilizumab

INTERVENTIONS:
Drug: CC-97540 — Specified dose on specified days
  Other Names: BMS-986353
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days
Drug: Tocilizumab — Specified dose on specified days

SUMMARY:
The purpose of this study is to establish the tolerability, preliminary efficacy, and pharmacokinetics of CC-97540 in participants with severe, refractory autoimmune diseases (Breakfree-1).

ELIGIBILITY:
Inclusion Criteria

- Diagnosis of Systemic Lupus Erythematosus (SLE) defined as follows:.

i) Fulfilling the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) classification criteria of SLE.

ii) Presence of anti-dsDNA, anti-histone, anti-chromatin, anti-Ro (anti-SS-A), anti-La (anti-SS-B), or anti-Sm antibodies at screening.

- SLE disease activity:.

i) Active disease at screening, with recent ≥ 1 major organ system with a BILAG A score (excluding musculoskeletal, mucocutaneous, and/or constitutional organ system).

ii) Inadequate response to glucocorticoids and to at least 2 of the following treatments, used for at least 3 months each: cyclophosphamide, mycophenolic acid or its derivatives, belimumab, azathioprine, anifrolumab, methotrexate, rituximab, obinutuzumab, cyclosporin, tacrolimus or voclosporin.

* Diagnosis of Idiopathic Inflammatory Myopathy (IIM) defined as follows:.

  i) Fulfilling the 2017 EULAR/ACR classification criteria for probable or definite IIM.

ii) Participant diagnosed with the following IIM subgroups: dermatomyositis (DM), immune-mediated necrotizing myopathy (IMNM), anti-synthetase syndrome (ASyS), and polymyositis (PM).

iii) Presence of at least 1 myositis specific antibody (MSA), associated antibody (MAA), or ANA at screening or prior to screening.

* IIM disease activity:.

  i) Severe/moderate muscle AND/OR skin involvement.

ii) Proof of activity as documented by:.

A. An active myositis-associated rash OR.

B. A recent muscle biopsy OR.

C. An elevated CK > 3 times the upper limit of normal OR.

D. Participants diagnosed IIM AND progressive Interstitial Lung Disease (ILD) on high-resolution computed tomography (HRCT)

iii) Inadequate response to glucocorticoids and at least 2 of the following treatments used for at least 3 months: azathioprine, methotrexate, cyclosporin A, tacrolimus, MMF, cyclophosphamide, IVIG, JAK inhibitors, and rituximab.

* Diagnosis of Systemic Sclerosis (SSc) defined as follows:.

  i) Fulfilling 2013 EULAR/ACR classification criteria for SSc.

ii) Antinuclear Antibody (ANA) positive at screening or prior to screening.

- SSc disease activity:.

i) Participants diagnosed with diffuse cutaneous SSc OR diffuse or limited cutaneous SSc AND progressive ILD, AND.

ii) Inadequate response to at least 1 of the following treatments used for at least 3 months: mycophenolate, cyclophosphamide, rituximab, nintedanib, azathioprine, tocilizumab, or intravenous immunoglobulins (IVIG).

- Rheumatoid Arthritis (RA) disease activity:.

i) Minimum of 3 SJC and 3 TJC on a 66/68 joint count (SJC/TJC).

ii) OR participants diagnosed with progressive ILD (interstitial lung disease).

iii) AND Inadequate disease response or intolerance to at least one conventional synthetic disease-modifying antirheumatic drug (DMARD) and as well as ≥ 2 DMARDs with different mechanisms of action from the categories biologic disease-modifying antirheumatic drug (bDMARDs) or targeted synthetic disease-modifying anti-rheumatic drug (tsDMARD) for a minimum of 3 months.

A. Participants qualifying on progressive ILD may have exhausted the therapies above OR have demonstrated inadequate disease response or intolerance to at least one of the following treatments used for at least 3 months: mycophenolate, tocilizumab, cyclophosphamide, rituximab, azathioprine, nintedinib, pirfenidone.

Exclusion Criteria

- Diagnosis of drug-induced SLE rather than idiopathic SLE.

- Other systemic autoimmune diseases (eg, multiple sclerosis, psoriasis, inflammatory bowel disease, etc) are excluded. Participants with type I autoimmune diabetes mellitus, thyroid autoimmune disease, Celiac disease, or secondary Sjögren's syndrome are not excluded.

* SLE overlap syndromes including, but not limited to, rheumatoid arthritis, scleroderma, and mixed connective tissue disease, are excluded.
* Present or recent clinically significant CNS pathology, within 12 months.
* IIM disease activity:.

  i) Other forms of IIM: Inclusion Body Myositis, Amyopathic DM, any form of juvenile myositis.

ii) Myositis other than IIM, eg, drug-induced myositis and PM associated with HIV.

iii) Participants with severe muscle damage (Physician VAS for muscle damage in Myositis Damage Index > 7 cm on a 10 cm scale), permanent weakness due to a non-IIM cause (eg, stroke), or myositis with cardiac involvement.

- SSc disease activity:.

i) SSc related PAH requiring active treatment.

ii) Rapidly progressive SSc related lower GI (small and large intestines) involvement (requiring parenteral nutrition); active gastric antral vascular ectasia.

iii) Prior scleroderma renal crisis.

- RA disease activity:.

i) Prior history of or current inflammatory joint disease other than RA.

ii) Joint damage and/or deformity that may confound the investigator's ability to accurately assess disease activity.

- Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2028-08-29 (Estimated); Study Completion 2028-08-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (AEs) in each indication. | Up to 2 years after CC-97540 infusion
Number of participants with serious AEs (SAEs) in each indication. | Up to 2 years after CC-97540 infusion
Number of participants with AEs of special interest (AESI) in each indication. | Up to 2 years after CC-97540 infusion
Number of participants with laboratory abnormalities in each indication. | Up to 2 years after CC-97540 infusion
Number of participants with Dose Limiting Toxicities (DLT) in each indication. | Up to 2 years after CC-97540 infusion
Recommended Phase 2 Dose (RP2D) of CC-97540 in each indication. | Up to 2 years after CC-97540 infusion

SECONDARY OUTCOMES:
Proportion of participants achieving definition of remission in SLE (DORIS) remission | At week 24
  SLE Cohort
Proportion of participants achieving Lupus Low Disease Activity State (LLDAS) | At week 24
  SLE Cohort
Change in proteinuria measured by urine protein creatinine ratio (UPCR) | At week 24
  SLE Cohort
Change in Health Assessment Questionnaire - Disability Index (HAQ-DI) | At week 24
Proportion of participants achieving Myositis Response Criteria (MRC) Total Improvement Score (TIS) Major Response | At Week 24
  IIM Cohort
Change in the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) | At Week 24
  Only Dermatomyositis (DM) participants in the IIM Cohort
Proportion of participants with ILD with no worsening of pulmonary function including forced expiratory volume (FEV1) (> 10%), forced vital capacity (FVC) (> 10%), and diffusing capacity of the lung for carbon monoxide (DLCO) (> 15%) | At Week 24
  IIM Cohort
Proportion of participants achieving a minimal clinically important difference (MCID) of 24% change from baseline of the modified Rodnan Skin Score (mRSS) | At Week 24
  SSc Cohort
Participants with an improvement from baseline of the Revised Composite Response Index in Systemic Sclerosis (CRISS) | At Week 24
  SSc Cohort
The worsening of pulmonary function including FVC (>10% absolute), DLCO (>15% absolute decline) in participants with interstitial lung disease (ILD) | At Week 24
  SSc Cohort
Proportion of participants achieving low Disease Activity Score-28 Joint C-Reactive Protein (DAS28-CRP) | At week 24
  RA cohort
Proportion of participants achieving simplified disease activity index (SDAI) remission | At week 24
  RA cohort
Proportion of participants with ILD with no worsening of pulmonary function including FVC (> 10%) | At week 24
  RA cohort
Maximum observed blood concentration (Cmax) | Up to 2 years
Time of maximum observed blood concentration (Tmax) | Up to 2 years
Area under the blood concentration-time curve from time zero to 28 days after dosing (AUC(0-28D)) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (30):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Local Institution - 0048, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Local Institution - 0053, Chicago, Illinois
  - Local Institution - 0030, Baltimore, Maryland
  - Local Institution - 0038, Boston, Massachusetts
  - Local Institution - 0046, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Local Institution - 0028, Omaha, Nebraska
  - Atlantic Health System Overlook Medical Center, Summit, New Jersey
  - NYU Langone Health, New York, New York
  - Local Institution - 0054, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Local Institution - 0055, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 0027, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
  - Local Institution - 0057, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium
- France (8):
  - Local Institution - 0043, Strasbourg, Alsace
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - CHU Montpellier Lapeyronie Hospital, Montpellier, Hérault
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Hôpital Saint-Louis, Paris
  - Local Institution - 0052, Paris
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
- Germany (7):
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité - Universitaetsmedizin Berlin - Campus Bejnamin Franklin, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Rome, Lazio
  - Humanitas, Rozzano, Milano
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario Reina Sofia, Córdoba
  - H.R.U Málaga - Hospital General, Málaga

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05869955.html